CLINICAL TRIAL: NCT00490516
Title: A Six-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Phase II Study of the Efficacy and Safety of ACP-104 in Acutely Psychotic Subjects With Schizophrenia
Brief Title: ACP-104 in Acutely Psychotic Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-104-003
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, psychotic disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: ACP-104
- 2 (Experimental)
  Interventions: Drug: ACP-104
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-104 — 200 mg, tablet, BID, 6 weeks
  Arms: 2
Drug: ACP-104 — 100 mg, tablet, BID, 6 weeks
  Arms: 1
Drug: Placebo — placebo, tablet BID, 6 weeks
  Arms: 3

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel-group, 6-week study, evaluating two dose levels of ACP-104 or Placebo twice a day in patients with schizophrenia who are experiencing an acute psychotic episode.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; 18-60 years of age
* The subject is physically healthy and medically stable.
* The subject is able to provide informed consent
* The subject has been diagnosed with schizophrenia for at least 1 year
* Currently experiencing an acute episode of psychosis
* The subject is willing to comply with all study-related events including in-patient hospitalization for at least 3 weeks.
* The subject has a caregiver who is willing and able to support the subject to ensure compliance with treatment and outpatient visits.
* If the subject is female, subject must be of non-childbearing potential - OR- if she is capable of becoming pregnant, agrees to commit to use one of the approved methods of contraception, as defined by the protocol.

Exclusion Criteria:

* If the subject is a pregnant or lactating (breast-feeding) female.
* The subject has a significant risk of suicide, homicide, and/or harm to self or others.
* Subject's psychotic symptoms have not improved with a therapeutic dose of antipsychotic treatment over the last 2 years.
* The subject is experiencing his/her first episode of schizophrenia.
* The subject has another psychotic disorder or has a history of autistic disorder or other pervasive developmental disorder (for example, mental retardation).
* The subject has been prescribed or exposed to clozapine before.
* The subject has donated blood or plasma within 56 days prior to the Screening Visit.
* The subject has participated in any clinical study within 30 days prior to the Screening Visit.

In addition to the criteria described above, subjects will be evaluated at screening to ensure that all criteria for study participation are met. These evaluations will include specific measures of the subject's health, including psychosis (mental health -the extent to which subject is unable to think clearly), heart condition, and pregnancy status. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline condition does not meet all protocol-specified entry criteria).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 247 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
PANSS | 6 weeks

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Anaheim, California
  - Costa Mesa, California
  - Covina, California
  - Culver City, California
  - Garden Grove, California
  - Glendale, California
  - Huntington Beach, California
  - Oceanside, California
  - Paramount, California
  - Pasadena, California
  - Pico Rivera, California
  - Riverside, California
  - San Diego, California
  - Bradenton, Florida
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Baltimore, Maryland
  - St Louis, Missouri
  - Willingboro, New Jersey
  - Philadelphia, Pennsylvania
  - Austin, Texas

IPD SHARING:
Plan to Share IPD: No